CLINICAL TRIAL: NCT00174733
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy of Ciclesonide Metered-Dose Inhaler at a Daily Dose of 160 μg Administered for Twelve Weeks Either in a Once-Daily Regimen in the Morning (160 μg qd AM) or in a Twice Daily Regimen (80 μg Bid) in Adults and Adolescents With Mild to Moderate Persistent Asthma Treated Previously With Inhaled Corticosteroids
Brief Title: Efficacy of Ciclesonide Versus Placebo Administered Either as Once Daily or Twice Daily in Patients Treated Previously With an Inhaled Corticosteroid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6163; XRP1526B/3030
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Asthma
Keywords: Glucocorticosteroid. Bronchospasm
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Ciclesonide (XRP1526)

SUMMARY:
To investigate the efficacy of ciclesonide MDI either as once daily or a twice daily regimen in patients with mild to moderate asthma, who have previously been treated with an inhaled corticosteroid.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 12 years or older
* History of persistent bronchial asthma for at least 6 months
* Documented use of an inhaled steroid or a combination of an inhaled steroid/long-acting beta 2 agonist for at least 1 month before screening
* At screening, FEV1 of 60 to 90% predicted or 70 to 95% predicted for either ICS or ICS/LABA use respectively.Reversibility of FEV1 by at least 12% and 200 ml post-bronchodilator
* Be able to use oral inhalers
* Non-smokers

Exclusion Criteria:

* History of life-threatening asthma
* Other pulmonary diseases; URI within 4 weeks before screening
* Use of systemic steroids within 1 month before screening or more than 3 times in previous 6 months
* Beta-adrenergic blocking agent use
* More than 2 in-patient hospitalizations or ER visits due to asthma exacerbations in the prior year before screening
* Pregnant or breast-feeding females
* Females of child-bearing potential not using adequate means of birth control
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease
* Abnormal clinical laboratory parameters that would limit participation in the study or interfere with interpretation of study results
* History of drug or alcohol abuse
* Treatment with any investigational product within 30 days prior to study entry

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2005-07; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 12 in FEV1

SECONDARY OUTCOMES:
Symptom scores, rescue albuterol use and morning peak flow measurements

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Meltzer EO, Korenblat PE, Weinstein SF, Noonan M, Karafilidis J. Efficacy and safety evaluation of ciclesonide in mild-to-moderate persistent asthma previously treated with inhaled corticosteroids. Allergy Asthma Proc. 2009 May-Jun;30(3):293-303. doi: 10.2500/aap.2009.30.3241. PMID 19549431